CLINICAL TRIAL: NCT00812643
Title: An Open, Single Centre Pharmacokinetic (Phase 1) Study of the Biliary Excretion of AZD0837 and Metabolites Following a Single Dose of [3H] AZD0837 Given in the Duodenum Via a Loc-I-Gut Catheter to Young Healthy Male Subjects
Brief Title: Excretion of Radiolabelled AZD0837
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Karin Wåhlander, MSD, AstraZeneca R&D Mölndal
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D1250C00032
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: pharmacokinetics
MeSH Terms: interventions — AZD 0837

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD0837 — Oral solution, dosing through the Loc-I-Gut catheter, single dose

SUMMARY:
This is an explorative study and the scientific question to be investigated in this study is if AZD0837 and/or its metabolites AR-H069927XX and AR-H067637XX and other unknown metabolites are excreted into the bile.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 19 to 30 kg/m2 and body weight between 50 to 100 kg inclusive

Exclusion Criteria:

* Significant illness, trauma or surgical procedures.
* Clinically significant laboratory abnormalities.
* Clinically significant medical history.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-01; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The amounts of total radioactivity excreted in bile. Metabolic profile of AZD0837 excreted in bile and identification of previously unknown metabolites and the amounts of AZD0837, AR-H069927XX and AR-H067637XX in bile. | Frequent sampling through a Loc-I-Gut catheter for up to 3 hours post dose.

SECONDARY OUTCOMES:
PK variables of AZD0837, AR-H069927XX, and AR-H067637XX. | Frequent sampling during 24 hours.
Adverse events, physical examination, safety laboratory variables, blood pressure, pulse and electrocardiography. | Some of the safety variables will be followed at each visit, some less frequent.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Knutson, MD, PhD, Principal Investigator — Inst för Kirurgiska VetenskaperUppsala Universitet
Locations (1):
- Research Site, Uppsala, Sweden